CLINICAL TRIAL: NCT01322919
Title: A Prospective Study to Evaluate the Safety and Effectiveness of the Presbyopic LASIK Algorithm
Brief Title: Safety and Efficacy Study to Evaluate the Treatment of Both Near and Distance Vision in a Simultaneous Laser Procedure
Acronym: Supracor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Myopia; Hyperopia; Presbyopia; Refractive Error
Keywords: PresbyLASIK; Presbyopia; LASIK; Supracor; refractive; Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia; Refractive Errors | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myopic Treatment Arm (Experimental): Patients treated in this arm will have preoperative measurements that indicate a myopic condition of the eye in conjunction with a presbyopic condition
  Interventions: Procedure: Supracor
- Hyperopic Treatment Arm (Experimental): Patients treated in this arm will have preoperative measurements that indicate a hyperopic condition of the eye in conjunction with a presbyopic condition
  Interventions: Procedure: Supracor

INTERVENTIONS:
Procedure: Supracor — All patients will undergo LASIK treatment on their non-dominant eye with a new laser software algorithm designed to treat both the distance and near vision components.
  The developed software algorithm uses the subjective refraction of the eye to create a treatment for the distance vision correction. This part of the treatment does not show any difference to a regular LASIK treatment for ametropic cases.
  In addition to the treatment for the distance vision a central ablation component will be added to address the near vision.
  Other Names: Myopia; Hyperopia; Presbyopia; PresbyLASIK; LASIK

SUMMARY:
By using a new software two consecutive laser treatments have been combined to correct the distance vision and to provide a near vision component in addition to the first treatment.

This study will help us to answer 2 questions:

1. How accurately this combined technique corrects distance and near vision
2. Whether the correction is adequate to remove the complete need for supplementary near spectacles

DETAILED DESCRIPTION:
LASIK is a surgical technique where the cornea is reshaped using a laser to provide visual correction. Typically, this procedure will only correct your long distance vision requiring the use of supplementary spectacles for reading and near vision.

The Technolas 217z Excimer Laser used to deliver the treatment is approved for use in the European Community for both treatment versions to correct separately the near vision and the distance vision for cases which need one or the other correction.

By using a new software two consecutive treatments have been combined to correct the distance vision and to provide a near vision component in addition to the first treatment.

This study will help us to answer 2 questions:

1. How accurately this combined technique corrects distance and near vision
2. Whether the correction is adequate to remove the complete need for supplementary near spectacles

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 45 years old and not older than 85 years
* Subjects must read, understand, and sign an Informed Consent Form (ICF).
* Subjects must be willing and able to return for scheduled follow up examinations through 6 months after surgery.
* Subjects must be willing to have both eyes treated with the laser during the same visit.
* Subjects for study arm-I must have up to +4 diopters (D) of absolute spherical hyperopia (not spherical equivalent), with up to +2.5 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction in both eyes. The spherical equivalent must be no more than +5.25 D. Subjects for study arm-II must have up to -7 diopters (D) of absolute spherical myopia (not spherical equivalent), with up to -4.0 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction in both eyes. The spherical equivalent must be no more than -9.00 D.
* Subjects must have presbyopia as determined by an age-related need for optical aid (> +1.50 D) for reading with their best distance correction.
* Subjects who have been screened successfully for acceptance of the PresbyLasik simulation
* Subjects who are contact lens wearers must have gas permeable (GP) lenses discontinued for at least 3 weeks and soft lenses discontinued for at least 1 week prior to the preoperative evaluation in the eye to be treated. Contact lens wearers who wear their contact lenses for any amount of time between the preoperative baseline examination and the operative visit must not be treated.
* Corneal topography should be normal.
* Subjects who are contact lens wearers must have 2 central keratometry readings and 2 manifest subjective refractions taken preoperatively at least one week apart. The refraction values must not differ by more than 0.50D as defined by manifest refraction spherical equivalent (MRSE). The keratometry values must not differ from the previous values by more than 0.50D in either meridian.
* High contrast, manifest, best spectacle-corrected logMAR distance visual acuity (VA) must be correctable to at least 0.1 (20/25 or 6/7.5) in both eyes.

Exclusion Criteria:

* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively.
* Eyes for which the baseline manifest subjective refraction exhibits a difference of greater than 0.75D in sphere power, or a difference of greater than 0.50D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than 0.75D, the difference in cylinder axis will not be taken into consideration.
* Subjects for whom the preoperative assessment of the ocular topography indicates that one or both eyes are not suitable candidates for treatment based upon the suggested computer-simulated treatment plan.
* Any subject who is going to be co-managed by an ophthalmologist or optometrist who is not approved as a Technolas Perfect Vision GmbH Excimer laser Investigator.
* Subjects with anterior segment pathology, including dry eye syndrome and cataracts which in the Investigator's opinion, would interfere with best spectacle-corrected VA (BSCVA) or a successful treatment.
* Subjects with evidence of retinal vascular disease.
* Subjects with any residual, recurrent, or active ocular disease, or corneal abnormality that in the Investigator's opinion would interfere with BSCVA or a successful treatment.
* Subjects with signs of keratoconus.
* Subjects with unstable central keratometry readings with irregular mires.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of excimer laser surgery for either refractive or therapeutic purposes.
* Subjects who have a history of Herpes simplex or Herpes zoster keratitis.
* Subjects who have a history of glaucoma or glaucoma suspect.
* Subjects who are immunocompromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, diabetes, autoimmune diseases and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Subjects taking systemic medications likely to affect wound healing such as corticosteroids or antimetabolites.
* Subjects who are known to be pregnant, lactating, or who plan to become pregnant during the course of the study.
* Subjects with known sensitivity to medications used for standard LASIK.
* Subjects participating in any other ophthalmic clinical trials during this clinical trial.
* Subjects with an ocular muscle disorder including a strabismus or nystagmus, or other disorders affecting fixation.
* Subjects at risk for angle closure.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The percentage of treated patients with an uncorrected monocular high contrast Near VA of 20/40 or better | 6 Months

SECONDARY OUTCOMES:
The percentage of treated eyes within +/- 1.00D of target refraction | 6 Months
The percentage of treated eyes within +/- 0.50D of target refraction | 6 Months
The percentage of treated eyes with a monocular uncorrected high contrast distance VA of 20/40 or better | 6 Months
Preservation of VA: Loss of more than 2 lines in monocular BCVA for distance vision | 6 Months
The percentage of treated eyes with an induced subjective manifest refraction cylinder not within +/- 2.00D | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Barragan, M.D., Principal Investigator — Laser Ocular Hidalgo
Locations (1):
- Laser Ocular Hidalgo, Monterrey, N.l., Mexico

REFERENCES:
- [Background] Telandro AP, Steile J 3rd. Presbyopia: perspective on the reality of pseudoaccommodation with LASIK. Ophthalmol Clin North Am. 2006 Mar;19(1):45-69, vi. doi: 10.1016/j.ohc.2005.10.006. PMID 16500528
- [Result] Epstein RL, Gurgos MA. Presbyopia treatment by monocular peripheral presbyLASIK. J Refract Surg. 2009 Jun;25(6):516-23. doi: 10.3928/1081597X-20090512-05. PMID 19603619
- [Result] Alio JL, Amparo F, Ortiz D, Moreno L. Corneal multifocality with excimer laser for presbyopia correction. Curr Opin Ophthalmol. 2009 Jul;20(4):264-71. doi: 10.1097/icu.0b013e32832a7ded. PMID 19537363
- [Result] Pinelli R, Ortiz D, Simonetto A, Bacchi C, Sala E, Alio JL. Correction of presbyopia in hyperopia with a center-distance, paracentral-near technique using the Technolas 217z platform. J Refract Surg. 2008 May;24(5):494-500. doi: 10.3928/1081597X-20080501-07. PMID 18494342
- [Result] Illueca C, Alio JL, Mas D, Ortiz D, Perez J, Espinosa J, Esperanza S. Pseudoaccommodation and visual acuity with Technovision presbyLASIK and a theoretical simulated Array multifocal intraocular lens. J Refract Surg. 2008 Apr;24(4):344-9. doi: 10.3928/1081597X-20080401-05. PMID 18500082
- [Result] Ortiz D, Alio JL, Illueca C, Mas D, Sala E, Perez J, Espinosa J. Optical analysis of presbyLASIK treatment by a light propagation algorithm. J Refract Surg. 2007 Jan;23(1):39-44. doi: 10.3928/1081-597X-20070101-07. PMID 17269242
- [Result] Alio JL, Chaubard JJ, Caliz A, Sala E, Patel S. Correction of presbyopia by technovision central multifocal LASIK (presbyLASIK). J Refract Surg. 2006 May;22(5):453-60. doi: 10.3928/1081-597X-20060501-06. PMID 16722483
- [Result] Becker KA, Jaksche A, Holz FG. [PresbyLASIK: treatment approaches with the excimer laser]. Ophthalmologe. 2006 Aug;103(8):667-72. doi: 10.1007/s00347-006-1391-y. German. PMID 16850290